CLINICAL TRIAL: NCT03195647
Title: PILOT STUDY for the Tight K TRIAL. Arrhythmias on the Cardiac Intensive Care Unit - Does Maintenance of High-normal Serum Potassium Levels Matter?
Brief Title: Pilot Study for the Tight K Study
Acronym: TightK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 011660
Record Dates: First submitted 2017-05-23; First posted 2017-06-22 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2018-06

CONDITIONS: Cardiac Arrythmias
Keywords: cardiovascular; potassium supplementation; coronary artery by pass surgery
MeSH Terms: interventions — Potassium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Relaxed control (Experimental): Those randomised to the 'Relaxed' Group will receive potassium supplementation only if their serum potassium drops below or equals 3.6 mEq/L.
  Interventions: Drug: Potassium
- Tight Control (Active Comparator): Patients randomised to the 'Tight' group will receive potassium supplementation if their serum potassium falls below 4.5 mEq/L (current practice).
  Interventions: Drug: Potassium

INTERVENTIONS:
Drug: Potassium — The trial treatment will start when patients are admitted to the intensive care unit after their surgery. The patient will undergo regular blood investigations, as per current practice. The frequency of K+ monitoring while on ICU will be according to clinician / nursing staff preference.
  Potassium supplementation will be according to local hospital protocols. This can be either via an intravenous infusion or as a tablet. Patients will otherwise be treated as per current hospital protocol.

SUMMARY:
The primary purpose of this pilot study will be feasibility of recruitment. However, in order to further inform a full randomised controlled trial (RCT), information on the incidence of atrial fibrillation (AF) and other arrhythmias, hospital length of stay, resource use and morbidity will be collected.

DETAILED DESCRIPTION:
Arrhythmias are common in critical care, with atrial tachyarrhythmias (and especially AF) being the most prevalent. This is especially true after cardiac surgery, with approximately 1 in 3 patients affected. The occurrence of new-onset post-operative AF is associated with increased short and long-term mortality, intensive care unit (ICU) and hospital stay and costs of care. This association appears causal, even after correction for confounding factors.

Potassium (K+) plays an important role in cardiac electrophysiology and abnormal levels may cause arrhythmias. Hypokalaemia, defined as a serum K+ <3.6 milliequivalents per litre (mEq/L) is thus associated with an increased incidence of ventricular arrhythmia after myocardial infarction. Low K+ levels are common following cardiac surgery, and appear marginally lower in those suffering atrial arrhythmias in this context. Despite an absence of proof that this association is causal, efforts to maintain serum [K+] in the 'high-normal' range (4.5 - 5.5 mEq/L) are considered 'routine practice' for AF prevention worldwide. The efficacy of such intervention remains unproven and data supporting this practice is extremely limited, being derived from observational rather than interventional studies. Indeed, no data exist to demonstrate that maintaining a high-normal potassium level is beneficial, or that aggressive replenishment of potassium in patients with heart disease necessarily leads to a better clinical outcome.

Furthermore, the method of potassium supplementation may be problematic. Oral replacement is not possible immediately post-operatively. Central venous administration is thus generally utilised in the early post-operative period. However, this practice is both time-consuming and costly: the intravenous administration of potassium carries recognised clinical risk, and is now prescribed in pre-diluted doses, stored securely for a safety purposes. Oral replacement is commonly associated with profound nausea, and is very poorly tolerated by patients. The investigators have estimated that the annual spending on potassium in cardiothoracic patients at Barts Health National Health Service (NHS) Trust is £100,000, compared to £16,500 for Milrinone (perceived as a high cost drug (2011-2012 prices). Additional costs relating to nursing time, drug checks, and intravenous connection and charting are also accrued. Central venous catheters may also be routinely left in situ solely for the purposes of parenteral potassium replacement; leading to an increased risk of line-related sepsis.

The routine maintenance of serum K+ in the high-normal range is thus a costly and unproven practice.

ELIGIBILITY:
Inclusion Criteria:

1. All patients undergoing isolated elective coronary artery bypass graft (CABG)

Exclusion Criteria:

1. Age less than 18 years
2. Previous AF
3. Concurrent patient involvement in another clinical study assessing post-operative interventions
4. On-going infection/sepsis at the time of operation
5. Pre-op high-degree atrioventricular (AV) block
6. Pre-op serum K+ greater than 5.5 mEq/L
7. Current or previous use of medication for the purposes of cardiac rhythm management
8. Dialysis dependent end stage renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Total number of patients recruited over a 6 month period | 6 months
  The pilot study is being conducted to assess if it is feasible to recruit the required patient population into the study. The aim of the pilot is to recruit 160 patients over 6 months from two different centres.
Number of patients successfully randomised into the study to receive standard either usual care or control of potassium at the lower limit of the normal range | 6 months
  The pilot study will investigate if it is feasible to randomised patients between the control and intervention arms of the study
Protocol violation rate | 6 months
  Feasibility of ensuring that protocol violation rate is no more than 10%
Number of patient with outcome data at 28 days | 6 months
  This is a feasibility and one of the main outcome will be to assess the number of participants with outcome data at 28 days. The study will aim to follow up 90% of the patients randomised.

SECONDARY OUTCOMES:
Incidence of new onset atrial fibrillation | Maximum of 5 days
  Episode of AF lasting at least 30 seconds that is clinically detected and/or electrocardiographically confirmed post surgery until day 5
Mean critical care length of stay | Maximum 28 days
  Average time patients are treated on critical care ward
Mean hospital length of stay | Maximum 28 days
  Average time patients are inpatients in all hospital wards
Incidence of all other arrhythmias, defined using standard diagnostic criteria | Maximum of 5 days
  All other arrhythmias detected clinically and/or review of holter monitor data
Incidence of in-patient mortality | 28 days from randomisation
  Number of patients deceased during their hospital stay
Incidence of mortality | 28 days from randomisation
  All incidence of mortality during hospital stay and follow up
Cost-effectiveness | 28 days from randomisation

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Barts Health NHS Trust, London
  - St George's University Hospital London, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Campbell NG, Allen E, Sanders J, Swinson R, Birch S, Sturgess J, Al-Subaie N, Elbourne D, Montgomery H, O'Brien B. The impact of maintaining serum potassium >/=3.6 mEq/L vs >/=4.5 mEq/L on the incidence of new-onset atrial fibrillation in the first 120 hours after isolated elective coronary artery bypass grafting - study protocol for a randomised feasibility trial for the proposed Tight K randomized non-inferiority trial. Trials. 2017 Dec 28;18(1):618. doi: 10.1186/s13063-017-2349-x. PMID 29282098